CLINICAL TRIAL: NCT02753582
Title: The Effect of Superoxide Dismutase (SOD) Enzyme on Frailty and Health Related Quality of Life Among Indonesian Pre-frail Elderly: A Double Blind Randomized Controlled Trial
Brief Title: The Effect of SOD Enzyme on Frailty and HRQOL Among Indonesian Pre-frail Elderly: A Double Blind Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Siti Setiati, Prof. MD, PhD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOD
Record Dates: First submitted 2016-04-12; First posted 2016-04-28 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Pre-frail Elderly
Keywords: Elderly, pre-frail, SOD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): SOD+Gliadin capsule is given in a dosage of 250 mg twice a day, for 24 weeks.
  Interventions: Dietary Supplement: SOD+Gliadin Capsule
- Placebo (Placebo Comparator): Placebo capsule is given in a dosage of 250 mg twice a day, for 24 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: SOD+Gliadin Capsule
  Other Names: GLISODin
  Arms: Intervention
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The primary objective is to determine the effect of SOD enzyme on frailty and health related quality of life among Indonesian pre-frail elderly.

The secondary objective is to determine the effect of SOD enzyme on anti-oxidant status, morbidity, and hospitalization among Indonesian pre-frail elderly.

The study hypothesis:

1. SOD enzyme can improve frailty status and health related quality of life among Indonesian pre-frail elderly.
2. SOD enzyme can increase anti-oxidant serum status among Indonesian pre-frail elderly.
3. SOD enzyme can decrease morbidity among Indonesian pre-frail elderly.
4. SOD enzyme can decrease hospitalization events among Indonesian pre-frail elderly.

DETAILED DESCRIPTION:
1. Study design: randomized double blind placebo controlled trial.
2. Location and time of study: Geriatric Outpatient Clinic and Internal Medicine Outpatient Clinic in Cipto Mangunkusumo National Hospital Jakarta. Study will be conducted on April 2016 to April 2017.
3. Study subject: elderly outpatient (aged 60 years old or more) with pre-frail status, who visit the clinic for medical consultation.
4. Data sampling: consecutive method.
5. Sample size: 150 subjects (75 control group, 75 intervention group).
6. Data collection: demographic data, frailty status, health related quality of life, anthropometric data, anti-oxidant serum status, hospitalization during intervention, morbidity, nutritional status, food intake, hand grip strength.
7. Intervention: SOD+Gliadin in capsule with a dose of 250 mg twice a day for 24 weeks will be given to intervention group, while placebo group will be given placebo capsule (amylum).

ELIGIBILITY:
Inclusion Criteria:

* Elderly aged 60 years or more with pre-frail condition
* Patients with SOD enzyme deficiency
* Willing to participate

Exclusion Criteria:

* Patients with cognitive function impairment (AMT score < 8)
* Patients with depression (Geriatric depression scale score >= 10)
* Patients with history of cirrhotic hepatic disease or severe hepatic disease
* Patients with kidney function impairment
* Patients with gluten allergy and derivative products
* Patients consume other antioxidant and omega-3 supplement

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-02 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Frailty status | 6 months (24 weeks)
  Measured by FI-40 item questionnaire.

SECONDARY OUTCOMES:
Health related quality of life | 6 months (24 weeks)
  Measured by EQ5D questionnaire.
Anti-oxidant serum status | 6 months (24 weeks)
  Measured by erythrocyte antioxidant enzymes activity, i.e. superoxide dismutase (SOD), catalase (CAT), glutathione peroxidase (GPX).
Morbidity | 6 months (24 weeks)
  Measured by Cumulative Illness Rating Score (CIRS).
Hospitalization | 6 months (24 weeks)
  Observed hospitalization event during the study

CONTACTS AND LOCATIONS:
Overall Officials: Siti Setiati, Prof, MD, PhD, Study Chair — Fakultas Kedokteran Universitas Indonesia; Purwita Wijaya Laksmi, MD, Study Director — Fakultas Kedokteran Universitas Indonesia; Kuntjoro Harimurti, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia; Rahmi Istanti, MARS, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Cipto Mangunkusumo National Hospital, Jakarta, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salomon JA, Wang H, Freeman MK, Vos T, Flaxman AD, Lopez AD, Murray CJ. Healthy life expectancy for 187 countries, 1990-2010: a systematic analysis for the Global Burden Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2144-62. doi: 10.1016/S0140-6736(12)61690-0. PMID 23245606
- [Background] Rodriguez-Manas L, Fried LP. Frailty in the clinical scenario. Lancet. 2015 Feb 14;385(9968):e7-e9. doi: 10.1016/S0140-6736(14)61595-6. Epub 2014 Nov 6. No abstract available. PMID 25468154
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Laksmi PW. Frailty syndrome: an emerging geriatric syndrome calling for its potential intervention. Acta Med Indones. 2014 Jul;46(3):173-4. No abstract available. PMID 25348178
- [Background] Setiati S, Harimurti K, Dewiasty E, Istanti R, Mupangati YM, Ngestiningsih D, Purwoko Y, Aryana IS, Kuswardhani RT, Pramantara ID, Apandi M, Dwipa L, Budiningsih F, Dinda R, Widajanti N, Siburian P, Sunarti S, Umar S, Jim E, Junaidi-Ar. Profile of food and nutrient intake among Indonesian elderly population and factors associated with energy intake: a multi-centre study. Acta Med Indones. 2013 Oct;45(4):265-74. PMID 24448330
- [Background] Setiati S. Vitamin D status among Indonesian elderly women living in institutionalized care units. Acta Med Indones. 2008 Apr;40(2):78-83. PMID 19054885
- [Background] Gill TM, Gahbauer EA, Allore HG, Han L. Transitions between frailty states among community-living older persons. Arch Intern Med. 2006 Feb 27;166(4):418-23. doi: 10.1001/archinte.166.4.418. PMID 16505261
- [Background] Sumantri S, Setiati S, Purnamasari D, Dewiasty E. Relationship between metformin and frailty syndrome in elderly people with type 2 diabetes. Acta Med Indones. 2014 Jul;46(3):183-8. PMID 25348180
- [Background] Wang CP, Lorenzo C, Espinoza SE. Frailty Attenuates the Impact of Metformin on Reducing Mortality in Older Adults with Type 2 Diabetes. J Endocrinol Diabetes Obes. 2014;2(2):1031. PMID 25506599
- [Background] Kobayashi S, Asakura K, Suga H, Sasaki S; Three-generation Study of Women on Diets and Health Study Groups. Inverse association between dietary habits with high total antioxidant capacity and prevalence of frailty among elderly Japanese women: a multicenter cross-sectional study. J Nutr Health Aging. 2014 Nov;18(9):827-39. doi: 10.1007/s12603-014-0478-4. PMID 25389961
- [Background] Cloarec M, Caillard P, Provost JC, Dever JM, Elbeze Y, Zamaria N. GliSODin, a vegetal sod with gliadin, as preventative agent vs. atherosclerosis, as confirmed with carotid ultrasound-B imaging. Eur Ann Allergy Clin Immunol. 2007 Feb;39(2):45-50. PMID 17441415
- [Background] Ensrud KE, Ewing SK, Taylor BC, Fink HA, Cawthon PM, Stone KL, Hillier TA, Cauley JA, Hochberg MC, Rodondi N, Tracy JK, Cummings SR. Comparison of 2 frailty indexes for prediction of falls, disability, fractures, and death in older women. Arch Intern Med. 2008 Feb 25;168(4):382-9. doi: 10.1001/archinternmed.2007.113. PMID 18299493
- [Background] Peng C, Wang X, Chen J, Jiao R, Wang L, Li YM, Zuo Y, Liu Y, Lei L, Ma KY, Huang Y, Chen ZY. Biology of ageing and role of dietary antioxidants. Biomed Res Int. 2014;2014:831841. doi: 10.1155/2014/831841. Epub 2014 Apr 3. PMID 24804252
- [Background] Bjelakovic G, Nikolova D, Gluud C. Meta-regression analyses, meta-analyses, and trial sequential analyses of the effects of supplementation with beta-carotene, vitamin A, and vitamin E singly or in different combinations on all-cause mortality: do we have evidence for lack of harm? PLoS One. 2013 Sep 6;8(9):e74558. doi: 10.1371/journal.pone.0074558. eCollection 2013. PMID 24040282
- [Background] Persson T, Popescu BO, Cedazo-Minguez A. Oxidative stress in Alzheimer's disease: why did antioxidant therapy fail? Oxid Med Cell Longev. 2014;2014:427318. doi: 10.1155/2014/427318. Epub 2014 Jan 5. PMID 24669288
- [Background] Flores-Mateo G, Carrillo-Santisteve P, Elosua R, Guallar E, Marrugat J, Bleys J, Covas MI. Antioxidant enzyme activity and coronary heart disease: meta-analyses of observational studies. Am J Epidemiol. 2009 Jul 15;170(2):135-47. doi: 10.1093/aje/kwp112. Epub 2009 May 22. PMID 19465742
- [Background] Laosa O, Alonso C, Castro M, Rodriguez-Manas L. Pharmaceutical interventions for frailty and sarcopenia. Curr Pharm Des. 2014;20(18):3068-82. doi: 10.2174/13816128113196660705. PMID 24079768